CLINICAL TRIAL: NCT04166838
Title: The Clinical Study of CD19 UCAR-T Cells in Patients With B-cell Acute Lymphoblastic Leukemia (B-ALL)
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Longyao Biotechnology Inc., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: V1.0
Record Dates: First submitted 2019-11-10; First posted 2019-11-18 (Actual); Last update posted 2019-11-18 (Actual); Status verified 2019-11

CONDITIONS: B-cell Acute Lymphoblastic Leukemia (B-ALL); Safety and Efficacy of CD19 UCAR-T Cells
MeSH Terms: conditions — Burkitt Lymphoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CD19 UCAR-T (Experimental)
  Interventions: Biological: CD19 UCARTcells

INTERVENTIONS:
Biological: CD19 UCARTcells — This study did not set up a control group. The maximum dose was determined according to the dose escalation test. Based on the number of CART cells per kg body weight which was proved to be safe and effective, all the subjects were treated with one single dose of CD19 UCART cells per treatment course. The dose escalation test was designed to evaluate the three dose levels of CD19 UCART (1 × 10 ^ 6 cells/kg,3 × 10 ^ 6 cells/kg,5 × 10 ^ 6 cells/kg). Each CD19 UCART infusion will be carried out on day 0. Each subject was observed for at least 4 weeks after the last infusion. If there was no dose-limited toxicity (DLT), it is necessary to continue multiple treatment courses at this dose level. The detailed administration time and dose were decided by the researchers.

SUMMARY:
This is a single arm, open-label, single center, exploratory clinical study to evaluate the safety and efficacy of CD19 UCAR-T Cells in Patients With CD19+ B-cell acute lymphoblastic leukemia (B-ALL).

DETAILED DESCRIPTION:
This study did not set up a control group. The maximum dose was determined according to the dose escalation test. Based on the number of CART cells per kg body weight which was proved to be safe and effective, all the subjects were treated with one single dose of CD19 UCART cells per treatment course. The dose escalation test was designed to evaluate the three dose levels of CD19 UCART (1 × 10 ^ 6 cells/kg,3 × 10 ^ 6 cells/kg,5 × 10 ^ 6 cells/kg). Each CD19 UCART infusion will be carried out on day 0. Each subject was observed for at least 4 weeks after the last infusion. If there was no dose-limited toxicity (DLT), it is necessary to continue multiple treatment courses at this dose level. The detailed administration time and dose were decided by the researchers.

ELIGIBILITY:
Inclusion Criteria:

* 1. Subjects between 6 and 70 years of age, inclusive.
* 2. Subjects diagnosed as relapsed or refractory B cell acute lymphocytic leukemia (B-ALL):

  1. Relapse as defined by 2nd or greater BM relapse or Any BM relapse after allogeneic SCT, naive lymphocytes in BM≥5%；
  2. refractory as defined by not achieving a CR after 2 rounds of standard chemotherapy.
* 3. Life expectancy > 12 weeks.
* 4. ECOG score between 0 and 1.
* 5. Liver, Renal, Heart and Lungs function defined as:

  1. Creatininec≤1.5 ULN;
  2. ALT/AST ≤2.5 ULN;
  3. Total Bilirubin≤1.5×ULN;
  4. Pulse oxygenation≥92%;
  5. Left Ventricular Shortening Fraction (LVSF)≥50%;
* 6. Subjects could comprehend the clinical study and able to provide written consent at the time of consent or assent.

Exclusion Criteria:

* 1. Pregnant or lactating women, or men or women with pregnancy plans within 6 months.
* 2. Subjects with contagious disease，such as HIV, active HBV and HCV, and syphilis, etc.
* 3. Subjects with mental or psychological illness who cannot be combined with treatment and efficacy evaluation.
* 4. Subjects with severe autoimmune disease and long-term use of immunosuppressants.
* 5. Subjects with active or uncontrollable infections requiring systemic treatment within 14 days prior to enrollment.
* 6. Subjects with any unstable systemic disease including, but not limited to, active infection (except for local infection), unstable angina pectoris, cerebrovascular accident or transient cerebral ischemia (within 6 months prior to screening), myocardial infarction (within 6 months prior to screening), congestive heart failure (New York Heart Association [NYHA] classification ≥ III).
* 7. subjects combined with dysfunction of vital organs such as lung, brain and kidney.
* 8. subjects that Participated in other similar clinical trials within 6 months.
* 9. subjects currently receiving treatment for other gene therapy.
* 10. subjects combined with graft versus host disease (GVHD).
* 11. Other subjects judged by the researchers to be unsuitable for admission to the study.

Ages: 6 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-11-08 (Estimated); Primary Completion 2019-11-08 (Estimated); Study Completion 2019-11-08 (Estimated)

PRIMARY OUTCOMES:
The Adverse events (AEs) | 24 weeks
  Number of Participants With Treatment-Related Adverse Events as Assessed by CTCAE v4.0
Graft-versus-Host Disease (GVHD) | 42 days
  Number of Participants with the GVHD by monitoring the epithelial cell damage in target organs including skin, liver, and gastrointestinal tract.
Expression of CD19 UCART cells | 2 years
  Expression of CD19 UCART cells detected by flow cytometry in blood and bone marrow.
Detection of CD19 UCART cells | 2 years
  Detection of CD19 UCART cells in blood, bone marrow by Quantitative Polymerase Chain Reaction (q-PCR).

SECONDARY OUTCOMES:
Overall Remission Rate (ORR) | 2 years
Complete Remission (CR) | 2 years
Disease Stabilization (SD) | 2 years
Disease Progression (PD) | 2 years
Overall survival (OS) | 2 years
Progression-free survival (PFS) | 2 years
Disease-free survival (DFS) | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Yi Yao, ph.D, Study Chair — Shanghai Longyao Bio-Tech Co., Ltd.
Locations (1):
- The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu, China